CLINICAL TRIAL: NCT07122739
Title: Reducing Spontaneous Recovery Using Functional Connectivity Based Real-time Functional Magnetic Resonance Imaging Neurofeedback Targeting the Memory Control Network
Brief Title: Neurofeedback to Reduce Spontaneous Recovery of Threat Expectancy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Princeton University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kenneth Norman, Huo Professor in Computational and Theoretical Neuroscience, Trustees of Princeton University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: P50MH136296-8441-33a; P50MH136296 (NIH)
Record Dates: First submitted 2025-08-01; First posted 2025-08-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are always blind to condition assignment. Because of the way that participants are assigned to the active vs. sham neurofeedback conditions, the investigator who is collecting the data will be aware of condition assignment for a small number of participants at the start and end of the study, but otherwise the investigator who is collecting the data will not be aware of condition assignment until after the participant has been run.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Neurofeedback (Experimental): Active neurofeedback will reinforce negative dlPFC-hippocampal functional connectivity, as this is expected to increase memory control ability.
  Interventions: Behavioral: Active Real-time fMRI Neurofeedback
- Control Neurofeedback (Sham Comparator): Participants in the control neurofeedback group will receive the same instructions as the experimental group, but will receive sham neurofeedback.
  Interventions: Behavioral: Sham Real-time fMRI neurofeedback

INTERVENTIONS:
Behavioral: Active Real-time fMRI Neurofeedback — Active neurofeedback to target a functional connection associated with increased memory control ability
  Arms: Active Neurofeedback
Behavioral: Sham Real-time fMRI neurofeedback — Sham neurofeedback
  Arms: Control Neurofeedback

SUMMARY:
This study tests the efficacy of a new behavioral intervention with the goal of reducing spontaneous recovery of threat expectancy in healthy adults. This real-time functional magnetic resonance imaging (fMRI) neurofeedback intervention delivers feedback based on a functional connection between the prefrontal cortex and the hippocampus.

DETAILED DESCRIPTION:
Exposure therapy remains the most effective evidence-based treatment for a variety of anxiety related disorders; however, fear often returns over time. Pavlovian conditioning and extinction serve as a laboratory model for threat learning and exposure therapy, respectively. Studies utilizing these tasks can help uncover why exposure therapy fails to prevent the return of fear in some individuals. Pilot data suggest that there are specific behavioral phenotypes that individuals exhibit during a test of spontaneous recovery following Pavlovian acquisition and extinction. Specifically, some participants exhibit high spontaneous recovery, despite previously extinguishing their responses. The investigators hypothesize that individuals that exhibit this behavioral phenotype are also individuals for whom exposure therapy would be ineffective. These distinct phenotypes are also associated with different forms of computational inference, as revealed by fitting latent-cause inference models to behavioral data. In the case of individuals that exhibit high spontaneous recovery, latent cause inference modeling suggests that these participants are reinstating a latent cause associated with initial threat learning, which was protected from updating by the formation of a new cause during extinction.

A separate line of work has focused on understanding the behavioral consequences and neural mechanisms of voluntary thought suppression, or inhibitory memory control. This is the process through which an individual can suppress a memory to reduce the influence that it has over future cognition and emotion. The neural mechanisms of retrieval inhibition are well known and involve top-down inhibition from the right dorsal-lateral prefrontal cortex (dlPFC) to the hippocampus.

Here, the investigators aim to test the hypothesis that memory control ability is related to latent cause inference during Pavlovian conditioning and extinction, and by extension is related to spontaneous recovery. The goal of this project is to causally test this hypothesis by using real-time fMRI to directly strengthen individuals' memory control ability. Real-time fMRI (rt-fMRI) neurofeedback is a powerful tool that allows participants to modulate their own neural activity based on external cues (akin to biofeedback). Here, the investigators will provide participants feedback designed to help them increase their memory control ability. Specifically, the investigators will give participants positive feedback whenever the investigators detect negative dlPFC-hippocampal functional connectivity, which is the putative neural signature of successful memory inhibition. A control group will also be included, which will involve the delivery of sham placebo neurofeedback. The investigators predict that, following rt-fMRI neurofeedback, participants who received active neurofeedback aimed at increasing memory control will exhibit lower spontaneous recovery in a Pavlovian conditioning task compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50
* No history of psychiatric disorders or neurological disorders affecting the central nervous system.
* Are not currently taking psychoactive medication or drugs of abuse.
* Must be eligible to enter an MRI (i.e., no permanent metal or medical implants)
* Normal color vision
* Right-handed
* Full reading and writing English comprehension
* Must exhibit spontaneous recovery behavior as determined by an experimenter in a prescreening experimental session
* Must be able to provide informed consent

Exclusion Criteria:

* Pregnancy (female participants)
* Outside of age range
* History of psychiatric or neurological disease
* Currently taking psychoactive medication or drugs of abuse
* Color blindness
* Primary left-handedness
* Less than full reading and writing English comprehension
* Do not exhibit spontaneous recovery behavior as determined by an experimenter in a prescreening experimental session
* Refusing to provide informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Spontaneous recovery behavior | Baseline and fourth fMRI session (out of four total fMRI sessions). At most 60 days will elapse between the start of data collection for a participant and their final fMRI session.
  The investigators will assess neurofeedback related changes in behavioral threat expectancy ratings in a discriminatory Pavlovian conditioning task. Spontaneous recovery is taken as the difference in responding to the conditioned stimulus that was paired with an outcome (CS+) vs. the conditioned stimulus that was not paired with an outcome (CS-) during a test of extinction recall following acquisition and extinction learning.

SECONDARY OUTCOMES:
Neurofeedback learning | Second and third fMRI sessions (out of four total fMRI sessions). At most 60 days will elapse between the start of data collection for a participant and their final fMRI session.
  The investigators will assess the overall trend in neurofeedback scores over the course of the intervention. If neurofeedback learning is successful, the investigators expect participants in the experimental group to increase the number of positive neurofeedback instances as the experiment progresses.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A. Norman, Ph.D., Principal Investigator — Princeton University
Locations (1):
- Princeton Neuroscience Institute, Princeton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be uploaded to the NIMH Data Archive (NDA).